CLINICAL TRIAL: NCT06146426
Title: Effects of Early Oral Diet After Cardiac Surgery: an Open Label Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MRC-01-23-507
Record Dates: First submitted 2023-11-19; First posted 2023-11-24 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-11

CONDITIONS: Adult Cardiac Surgery

STUDY DESIGN:
Intervention Model Description: This is an open label randomized controlled trial with two parallel groups. No blinding will be considered.Patients will be randomly assigned to either early or conventional oral feeding group using software STATA 17.0 or SPSS 24.0. Sequentially numbered opaque sealed envelopes (SNOSE) which contain the allocation will be used. These envelopes are prepared by an independent person who is not a research team member. It will be sealed and provided to the principal investigator or co-investigator or statistician.Subjects will be enrolled as per the inclusion criteria. The patients will be approached directly in the preoperative period and informed consent will be obtained.
  They will be allocated to early and conventional diet groups by randomization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early diet (Experimental): The patients of early group will be performed water swallowing test at bedside after 2 hours of extubation. Before performing the Water Swallow Test, the patient must be evaluated for readiness.This interventional group of patients will be initiated with sips of water (warm or cold as patient prefers) at 2 hours of extubation (post-operative day 0) followed by clear liquid diet (tea, clear juice/ soup, gelatin) at 4 hours. If well tolerated, then slowly progress to a full liquid and solid diet as the patient preferred pace.
  Interventions: Dietary Supplement: Early diet resumption
- Conventional diet (No Intervention): Patients in this group will receive the existing standard (conventional) post-operative diet regimen that is sips of water on the day of surgery and initiation of solid oral diet on next day (post-operative day 1)

INTERVENTIONS:
Dietary Supplement: Early diet resumption — Resuming oral diet at pace started from 2 hours after extubation from ventilator.
  Arms: Early diet

SUMMARY:
This is an open label randomized controlled trial with two parallel groups to compare the effects of early initiation of oral diet to reduce the post-operative fasting time in adult patients undergoing cardiac surgery.Primary Objectives:

* To assess the impact of early and conventional diet on post-operative nausea and vomiting by calculating the simplified PONV (post-operative nausea and vomiting) impact score of patients after cardiac surgery, with a score >5 indicating clinically significant PONV.
* To study the impact of early versus conventional diet on gastrointestinal function by estimating the difference in timing of the first bowel movement in patients following cardiac surgery.

Secondary Objectives:

* To evaluate the effects of early versus conventional diet resumption on length of ICU stay among the patients following cardiac surgery in days.
* To compare the satisfaction levels of patients by visual analogue scale who resumed their oral diets early versus conventionally following cardiac surgery. The estimated sample size of 196 patients with routine post operative recovery after cardiac surgery will be randomized into early (interventional) and late (control) diet groups. Researchers will compare the early diet group with late diet group to see the effects.

DETAILED DESCRIPTION:
This is an open label randomized controlled trial with two parallel groups to compare the effects of early initiation of oral diet to reduce the post-operative fasting time in adult patients undergoing cardiac surgery. Assuming a incidence rate of post-operative nausea and vomiting of 40% in cardiac surgery (Sawatzky et al., 2014), and an anticipated incidence of clinically significant PONV using the simplified PONV impact scale of 20% (Myles et al., 2012), with a presumed 50% risk reduction with early feeding, a power of 80%, and alpha of 0.05, the minimum effective sample size would be 164 subjects (82 per arm). Assuming a drop out of 20%, the sample size was increased to 196 subjects (98 per arm).

Adult patients' status post-operative cardiac surgery in CTICU of Heart Hospital, after extubation, meeting inclusion criteria will be included in the study.

They will be divided into early and conventional diet groups. and randomized using web-based randomization to early diet (intervention arm) versus conventional diet (control arm) in 1:1 ratio. The patients of early group will be examined for water swallowing test (WST) at bedside after extubation. Before performing the WST, the patient must be evaluated for readiness including Awake, alert, cooperative, able to follow command, vital signs are stable, able to maintain at least 75-degree.

in upright position, the patient can cough effectively, the patient can stick out tongue and move to the left and right, the patient can breathe comfortable.

The patient's mouth will be cleaned, and the patient will be asked to drink each 5 ml of water (1 teaspoon) 3 times respectively. If the patient shows any abnormal signs, the test will be discontinued. If all steps are passed, then the patient will continue to drink the entire 90 ml of water from a cup or with a straw in sequential slowly and steadily swallowing without stopping (cup or straw can be held by clinician or patient). (Phothikun N, 2022).

If the patient fails in water swallow test, early diet will not be resumed. The finding will be intimated to the physician in charge of the patient for further management.

For the early group if they pass water swallow test oral diet will be resumed after 2 hours of extubation with water, followed by clear liquid diet after 4 hours and gradually laddered to solid diet as patient prefers/tolerates. For the conventional diet group, the existing standard feeding protocol will be followed, that is patient will be given only sips of water on the day of surgery and the diet will be resumed on the next day after surgery.

The simplified post-operative nausea -vomiting impact score every 4th hourly for 24 hours, time of first bowel movement, the length of ICU stays in days and patient satisfaction level about timing of resuming oral diet using Visual analogue scale at the time of discharge from hospital (VAS) (Appendix 3) will be collected. Participants will be provided with VAS with a statement explaining what the scale was intended to measure that is the level of satisfaction on resuming diet early. Other signs of regaining gut functions like bowel sounds and flatus is not considered in this study because assessment of bowel sounds is not a reliable sign of gut function (Deane et.al,2021) and chances for ambiguity are high while the assessment of bowel sounds. Most of the patients after major surgery with general anaesthesia may not recognize the first flatus in immediate post-operative period. For the patient who is not tolerating the oral diet resumption with any signs of aspiration or clinically significant vomiting or paralytic ileus or patient dissatisfaction with oral diet resumption, early diet trial will be discontinued and reported accordingly.

The study will be conducted at a single center and the patients will be followed for 5 days after surgery. The favorable circumstances enhance safety of early resumption of oral diet in adult cardiac surgery are as follows. The short acting Propofol is used as the major sedation after surgery to prevent prolonged sedative effect. Multimodal analgesia is used to reduce the use of narcotics. Patient controlled analgesia of low dose morphine or fentanyl is used along with intravenous paracetamol and non-pharmacological interventions like massage, changing positions and early mobilization out of bed. Sedation score is assessed every hour by the intensive care nurses using Ramsay Sedation scale. All patients are routinely placed on intravenous metoclopramide injections as prokinetic and antiemetic which may help to enhance peristalsis. Patients are also given oral mucosal massage with flavored glycerin swab sticks to enhance their appetite.

All data will be analyzed using SPSS 24.0 statistical package. Descriptive statistics will be used to describe and compare socio-demographic data on participants between the intervention and control group. Continuous variables that follow a normal distribution will be expressed as means and standard deviations, whereas categorical variables will be presented as frequency counts and percentages. We will estimate simplified PONV (post-operative nausea vomiting) impact score for early and conventional diet groups. Quantitative data between the intervention and control groups will be analyzed using unpaired t or Mann Whitney U test as appropriate. Categorical data will be summarized using frequencies and proportions. Associations between two or more qualitative data variables will be assessed using Chi-square (χ2) test or Fisher Exact test as appropriate. Univariate and multiple regression analysis will be used to control and adjust for potential predictors and confounders such as type of age, gender, nationality and presence of comorbidities and motion sickness. Generalized estimating equation will be used to see the change over the post-operative nausea- vomiting impact score in both the groups over 24 hours. All tests will be two sided and p value considered <0.05 as significant.

No adverse events are expected in either of the groups. Any accidental adverse event will be reported immediately to the physician and the details of the event, harm and treatments will be notified to MRC. And the instructions by MRC will be followed. A record of such events will be maintained for further reference. This is to state that this study will be conducted in full conformance with principles of the "Declaration of Helsinki", Good Clinical Practice (GCP) and within the laws and regulations of MoPH in Qatar. The participants will be able to withdraw from the study anytime without any liabilities during the research process.

ELIGIBILITY:
Inclusion Criteria:

* Patients' post-operative status,
* Post extubation (usually extubated within 4-6 hours after surgery) without any cognitive deficits, expected
* Minimal chest drain (<100 ml/h), with
* Awake, alert, oriented without any cognitive impairment
* Able to pass water swallow test will be included in the study.

Exclusion Criteria

* Major complicated cardiac surgeries (aortic dissection, surgeries involving mechanical circulatory support (ECMO or Ventricular assist devices).
* Patients with profuse surgical /chest drain bleeding >100 ml/h for 3 consecutive hours in chest drain,
* Patients undergo re-exploration sternotomy, cardiac tamponade and
* Patients with cognitive impairment, drowsy
* Absence of vocalization after extubation
* Patients who fails in water swallow test for dysphagia after extubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
simplified post operative nausea vomiting impact score. | 24 hours
  To assess the impact of early and conventional diet on post-operative nausea and vomiting by calculating the simplified PONV (post-operative nausea and vomiting) impact score of patients after cardiac surgery, with a score >5 indicating clinically significant PONV.
Timing of bowel movements | 5 days
  To study the impact of early versus conventional diet on gastrointestinal function by estimating the difference in timing of the first bowel movement in patients of both groups following cardiac surgery.

SECONDARY OUTCOMES:
length of ICU stays in days. | 5 days
  To evaluate the effects of early versus conventional diet resumption on length of ICU stay among the patients following cardiac surgery in days.
patient satisfaction | 2 days
  To compare the satisfaction levels of patients by visual analogue scale who resumed their oral diets early versus conventionally. Visual analogue scale scores range from 1 to 5 where 1 indicates extremely dissatisfied with early diet resumption and 5 indicates extremely satisfied.
  following cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Siddiha P Shahulhameed, Principal Investigator — Hamad Medical Corporation
Locations (1):
- Heart Hospital, Doha, Qatar

REFERENCES:
- [Background] Bowling TE. Does disorder of gastrointestinal motility affect food intake in the post-surgical patient? Proc Nutr Soc. 1994 Mar;53(1):151-7. doi: 10.1079/pns19940018. PMID 8029224
- [Background] Brown JK, Singh K, Dumitru R, Chan E, Kim MP. The Benefits of Enhanced Recovery After Surgery Programs and Their Application in Cardiothoracic Surgery. Methodist Debakey Cardiovasc J. 2018 Apr-Jun;14(2):77-88. doi: 10.14797/mdcj-14-2-77. PMID 29977464
- [Background] Charoenkwan K, Phillipson G, Vutyavanich T. Early versus delayed (traditional) oral fluids and food for reducing complications after major abdominal gynaecologic surgery. Cochrane Database Syst Rev. 2007 Oct 17;(4):CD004508. doi: 10.1002/14651858.CD004508.pub3. PMID 17943817
- [Background] Feng S, Chen L, Wang G, Chen A, Qiu Y. Early oral intake after intra-abdominal gynecological oncology surgery. Cancer Nurs. 2008 May-Jun;31(3):209-13. doi: 10.1097/01.NCC.0000305729.57722.a7. PMID 18453877
- [Background] Hill A, Nesterova E, Lomivorotov V, Efremov S, Goetzenich A, Benstoem C, Zamyatin M, Chourdakis M, Heyland D, Stoppe C. Current Evidence about Nutrition Support in Cardiac Surgery Patients-What Do We Know? Nutrients. 2018 May 11;10(5):597. doi: 10.3390/nu10050597. PMID 29751629
- [Background] Jejurikar SS, Orseck MJ, Matarasso A. Reevaluating resumption of oral intake after abdominoplasty. Aesthet Surg J. 2007 May-Jun;27(3):233-8. doi: 10.1016/j.asj.2007.03.004. PMID 19341649
- [Background] Kolodziej T, Maciejewski T, Mendrala K, Darocha T, Weglarzy A, Budziarz B, Kiermasz K, Kucewicz-Czech EM. Enhanced recovery after cardiac surgery. Kardiochir Torakochirurgia Pol. 2019 Mar;16(1):32-36. doi: 10.5114/kitp.2019.83943. Epub 2019 Apr 4. PMID 31043973
- [Background] Minig L, Biffi R, Zanagnolo V, Attanasio A, Beltrami C, Bocciolone L, Botteri E, Colombo N, Iodice S, Landoni F, Peiretti M, Roviglione G, Maggioni A. Reduction of postoperative complication rate with the use of early oral feeding in gynecologic oncologic patients undergoing a major surgery: a randomized controlled trial. Ann Surg Oncol. 2009 Nov;16(11):3101-10. doi: 10.1245/s10434-009-0681-4. PMID 19760046
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Ogbadua AO, Agida TE, Akaba GO, Akitoye OA, Ekele BA. Early Versus Delayed Oral Feeding after Uncomplicated Cesarean Section under Spinal Anesthesia: A Randomized Controlled Trial. Niger J Surg. 2018 Jan-Jun;24(1):6-11. doi: 10.4103/njs.NJS_26_17. PMID 29643726
- [Background] Osland E, Yunus R, Khan S, Memon MA. Early enteral nutrition within 24 h of intestinal surgery versus later commencement of feeding: a systematic review and meta-analysis. J Gastrointest Surg. 2009 Jun;13(6):1163-5; author reply 1166-7. doi: 10.1007/s11605-009-0846-2. Epub 2009 Mar 6. No abstract available. PMID 19266244
- [Background] Stoppe C, Goetzenich A, Whitman G, Ohkuma R, Brown T, Hatzakorzian R, Kristof A, Meybohm P, Mechanick J, Evans A, Yeh D, McDonald B, Chourdakis M, Jones P, Barton R, Tripathi R, Elke G, Liakopoulos O, Agarwala R, Lomivorotov V, Nesterova E, Marx G, Benstoem C, Lemieux M, Heyland DK. Role of nutrition support in adult cardiac surgery: a consensus statement from an International Multidisciplinary Expert Group on Nutrition in Cardiac Surgery. Crit Care. 2017 Jun 5;21(1):131. doi: 10.1186/s13054-017-1690-5. PMID 28583157
- [Background] Stoppe C, Whitlock R, Arora RC, Heyland DK. Nutrition support in cardiac surgery patients: Be calm and feed on! J Thorac Cardiovasc Surg. 2019 Oct;158(4):1103-1108. doi: 10.1016/j.jtcvs.2019.02.132. Epub 2019 May 7. No abstract available. PMID 31202453
- [Background] Tatsuishi W, Kohri T, Kodera K, Asano R, Kataoka G, Kubota S, Nakano K. Usefulness of an enhanced recovery after surgery protocol for perioperative management following open repair of an abdominal aortic aneurysm. Surg Today. 2012 Dec;42(12):1195-200. doi: 10.1007/s00595-012-0252-3. Epub 2012 Jul 14. PMID 22797961
- [Background] Visser M, Davids M, Verberne HJ, Kok WE, Tepaske R, Cocchieri R, Kemper EM, Teerlink T, Jonker MA, Wisselink W, de Mol BA, van Leeuwen PA. Nutrition before, during, and after surgery increases the arginine:asymmetric dimethylarginine ratio and relates to improved myocardial glucose metabolism: a randomized controlled trial. Am J Clin Nutr. 2014 Jun;99(6):1440-9. doi: 10.3945/ajcn.113.075473. Epub 2014 Apr 2. PMID 24695897
- [Background] Voutilainen A, Pitkaaho T, Kvist T, Vehvilainen-Julkunen K. How to ask about patient satisfaction? The visual analogue scale is less vulnerable to confounding factors and ceiling effect than a symmetric Likert scale. J Adv Nurs. 2016 Apr;72(4):946-57. doi: 10.1111/jan.12875. Epub 2015 Dec 22. PMID 26689434
- [Background] Deane AM, Ali Abdelhamid Y, Plummer MP, Fetterplace K, Moore C, Reintam Blaser A. Are Classic Bedside Exam Findings Required to Initiate Enteral Nutrition in Critically Ill Patients: Emphasis on Bowel Sounds and Abdominal Distension. Nutr Clin Pract. 2021 Feb;36(1):67-75. doi: 10.1002/ncp.10610. Epub 2020 Dec 9. PMID 33296117
- [Background] Bours GJ, Speyer R, Lemmens J, Limburg M, de Wit R. Bedside screening tests vs. videofluoroscopy or fibreoptic endoscopic evaluation of swallowing to detect dysphagia in patients with neurological disorders: systematic review. J Adv Nurs. 2009 Mar;65(3):477-93. doi: 10.1111/j.1365-2648.2008.04915.x. PMID 19222645
- [Background] Phothikun, N., Thitisakulchai, P., Tanvijit, P., & Yuyen, T. (2022). The incidence and risk factors of post-extubation dysphagia in critically ill surgical patients: protocol for prospective observational study. Clinical Critical Care, 30. https://doi.org/10.54205/ccc.v30.254965